CLINICAL TRIAL: NCT06727292
Title: Biometrical Evaluation of the Efficacy of a Food Supplement Versus Placebo
Acronym: FB_BfW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Finzelberg GmbH & Co. KG (Industry)
Collaborators: Eurofins (Industry); Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUX824AA0245
Record Dates: First submitted 2024-11-26; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Skin Aging; Hair Condition; Skin Condition
Keywords: improvements of skin physiological parameters
MeSH Terms: conditions — Skin Diseases | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: single-center, ,double-blind, randomized pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the product is also masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo has similar characteristics as the verum instant drink.
  Interventions: Dietary Supplement: Placebo
- Food supplement (Experimental): Powder for an instant drink preparation with orange flavor /taste
  Interventions: Dietary Supplement: Food supplement

INTERVENTIONS:
Dietary Supplement: Food supplement — Instant drink in a powder form presented in a sachet to be disolved in a glass of water (200 ml).
  Arms: Food supplement
Dietary Supplement: Placebo — Instant drink in powder form in a sachet to be disolved in a glass of water (200ml)
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to evaluate whether nutritional supplementation over a 2-month period improves skin physiological parameters. This is a national, single-center, double-blind, randomized pilot study.

The study will be conducted using a supplement and a placebo, the safety of which has been assured by the sponsor.

Participants will:

* Take a food supplement or a placebo once daily for 2 months
* Visit the study center at beginning, after 28 days and after 56 days of supplementation.
* Keep a diary of their skin status and tolerability

The secondary objective is to evaluate product characteristics and performance during normal use in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Phototype: I to IV;
* Subjects with normal to dry skin;
* Subjects with healthy skin on the study area;
* Non-smokers;
* Has normal nutritional habits (not vegetarian/vegan);
* Is not pregnant or lactating;
* Has a BMI of 18 - 33 kg/m2;
* Is willing to refrain from taking dietary supplements (at best not at all, in any case not during the last month before study start);
* Willing not to use any oral products or any nutritional supplementation aiming at improving skin status during the course of the study;
* No history of malabsorption diseases, liver diseases, or diseases of the lipid metabolism;
* Uses no medication, which may interact with the study product

Exclusion Criteria:

* For women: pregnant or nursing woman or woman planning to get pregnant during the study;
* Cutaneous pathology on the study zone (eczema, etc.);
* Subject with make-up on the day of the visit at the laboratory;
* Use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the efficacy of the study product:

  * change in anti-wrinkle, smoothing and/or firming topical products within previous week on the studied zones,
  * non-invasive procedures within previous month on the studied zones,
  * intake of food supplement acting on skin within the three previous months,
  * invasive procedures:

    * deep chemical peeling within previous 3 months on the studied zones,
    * mesotherapy, dermapen, laser within previous 6 months on the studied zones,
    * botox and/or hyaluronic acid injections within previous 12 months on the studied zones;
* Intake of vitamin substances and diets comprising a change of normal eating habits;
* Known allergy to one or several investigational product´s ingredients;
* Participation in a nutritional study within the last 30 days;
* Surgical or internal diseases e.g. a metabolic or endocrine disease that may affect the outcome of the study (e.g. diabetes, liver diseases, kidney disorders) or having a history of medical or surgical events that may significantly affect the study outcome including any cardiovascular disease, skin disease, hypertension (>140/90 mm Hg in three repeated measurements).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 66 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Skin Physiological Parameters | Skin physiological parameters will be assessed at Day 0, Day 28, Day 56
  Changes in skin hydration: Measurement of skin hydration by means of a Corneometer CM825.
Skin Physiological Parameters | Skin physiological parameters will be assessed at Day 0, Day 28, Day 56
  Assessment of skin barrier integrity measuring transepidermal water loss using the Tewameter® TM 300.
Skin Physiological Parameters | Skin physiological parameters will be assessed at Day 0, Day 28, Day 56
  Change in skin elasticity using Cutometer MPA580
Skin Physiological Parameters | Skin physiological parameters will be assessed at Day 0, Day 28, Day 56
  Changes in skin density using ultrasound measurements with a frequency of 20 MHz (Derma Scan C, Vers. 3) with 2-D-configuration (Cortex Technology, Denmark).

SECONDARY OUTCOMES:
Subject satisfaction | It will be assessed at Day 28, Day 56
  A subjective evaluation questionnaire on the study product's effects on the skin will be completed by subjects (each item is scored individually on a 5 point Likert scale ranging from 'Totally agree' to 'Totally disagree')
Adverse events | Adverse events will be assessed during the whole study from Day 0 to Day 56
  Collection of adverse events throughout the study
Subject self-assessment quality of the skin and hair. | It will be assessed at Day 28, Day 56
  The quality of the volunteers' skin and hair will be subjectively assessed by a self-assessment questionnaire. This questionnaire will assess the volunteers' perception of improvement in their skin in general and in wrinkles, spots, redness, elasticity, hydration, appearance. In the case of hair, the questionnaire will assess if it is stronger than before. There will be 5 levels in the questionnaire to assess how true the statements are: No Information (0), No improvement (1), Somewhat (2), Clearly Yes (3) and Yes, Very clearly (4).

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Poland, Gdansk, GDANSK, Poland

IPD SHARING:
Plan to Share IPD: No
To comply with European regulations and national provisions, subjects are informed that not sharing of IPD is planned in order to protect their personal data. If data is to be shared, participants must be informed individually, and their consent obtained.